CLINICAL TRIAL: NCT05194891
Title: Specular Microscopic Changes of Corneal Endothelial Cells After Phacoemulsification in Patients With Pseudo Exfoliation
Brief Title: Endothelial Changes in Pseudoexfoliation Syndrome
Acronym: PEX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shymaa Ahmed, Principal Investigator, Assiut University
Other Study IDs: Endothelial Changes in PEX
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Endothelial Cell Loss, Corneal
MeSH Terms: conditions — Corneal Endothelial Cell Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Specular Microscopy — Phacoemulsification

SUMMARY:
this study aimed to evaluate the corneal endothelial cell changes before and after phacoemulsification in pseudoexfoliative patients relative to healthy adults.

DETAILED DESCRIPTION:
Pseudoexfoliation syndrome (PEX) is an age related microfibrillopathy disorder characterized by the deposition of greyish white flaky exfoliative material in ocular and extraocular tissue. It commonly affects patients over 50 years old ((commonly in late 60s and 70s) with prevalence range from 0.5% to > 30%, Although it occurs in virtually every area of the world, a considerable racial variation exists in its incidence. It is relatively rare among African Americans and Eskimos. Prevalence is high in the Sami people who are indigenous of northern Europe. There is also a high prevalence in Arabic populations. It is also well known that patients with PXF develop cataracts early in their lives. Phacoemulsification is a preferred type of cataract surgery owing to fewer complications than other types. However, it still has significant undesirable hazardous as Posterior capsular rupture, vitreous loss, Retinal detachment, Cystoid macular oedema and Posterior capsule opacification. Also, it can enhance loss of corneal endothelial cells, thickness and density that may result in corneal decompensation and subsequent corneal transplantation. In patients with PXF, small pupils and weak zonular support may enhance Phacoemulsification complications. Non-contact Specular microscope is a non-invasive method for morphological analysis of corneal density of endothelial cells, "size change" (Polymegathism), "hexagonal change" (pleomorphism). Therefore, this technology plays an important role in preoperative evaluation, surgical design and postoperative care.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is above50 years.
2. Patient with nuclear cataract grade II, III.
3. Clear cornea with no evidence of endothelial disease.
4. Endothelial cell density more than 1000\mm2.
5. Normal anterior chamber depth and dilatable pupil.
6. No active ocular disease or inflammation.
7. Pseudoexfoliative patients.

Exclusion Criteria:

1. History of previous trauma, intraocular surgery or ocular surface infection in recent two weeks.
2. Presence of any corneal opacity, endothelial disease, scarring or dystrophies.
3. Pseudoexfoliative glaucoma.
4. Patients age below 50 years.
5. Endothelial cell count less than 1000\mm2.

Ages: 50 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This prospective, non-randomized comparative ,interventional study was performed on 100 eyes of 100 patients who were divided equally into two groups (pseudoexfoliative and control). Patient who aged above50 years and with nuclear cataract grade II,III, clear cornea and endothelial cell density more than 1000\mm2 were included in this study. Also, patients with normal anterior chamber depth, dilatable pupil and with no active ocular disease or inflammation were included. Pseudoexfoliative patients who had glaucoma were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Study of corneal endothelial changes in pseudoexfoliation syndrome | Baseline
  Comparison of corneal endothelial changes after phacoemulsification in patients with pseudoexfoliation and patient with cataract only

CONTACTS AND LOCATIONS:
Overall Officials: Shymaa Sabet, Doctor, Principal Investigator — Assiut University